CLINICAL TRIAL: NCT01735734
Title: An Observational Study as to the Effects of Cutaneous Air-cooling on Blood Vessel Diameter in Capillary Malformations
Brief Title: Assessing the Effects of Air-cooling on Capillary Malformations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr Irving Ling, Academic Foundation Doctor, Honorary Clinical Fellow, NHS Greater Glasgow and Clyde
Other Study IDs: GN
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Capillary Malformation; Laser; Skin Cooling
Keywords: Skin disease; Capillary Malformation; Laser therapy
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Skin Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Capillary malformation
  Interventions: Device: Air cooling to CM site

INTERVENTIONS:
Device: Air cooling to CM site

SUMMARY:
The purpose of this observational study is to ascertain the effects of cutaneous air cooling on vessel diameter within Capillary Malformations (CM).

DETAILED DESCRIPTION:
Capillary malformation (CM) is the most common vascular malformation occurring in approximately 0.3% of all newborn. The standard treatment for facial or aesthetically sensitive CM's is flashlamp Pulsed Dye Laser. Skin cooling prior to laser treatment of CMs is standard practice within our department. The effects of skin cooling on the vasculature within CMs are poorly understood. Previous studies by our department have shown that raising ambient temperature increases CM vessel size. It has been postulated that by increasing CM vessel size, it may also increase the effectiveness of treatment. We hypothesize that cooling the skin during laser treatment may cause vasconstriction of the superficial vessels within the CM. This may have an impact on treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Adult more than 16 years of age
* Patient diagnosed with Capillary Malformation

Exclusion Criteria:

* Patients less than 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Capillary Malformation identified through our department database
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
To study the effects of cutaneous air cooling on blood vessel diameter in capillary malformation | 10 minutes
  In a temperature controlled room, the participant's capillary diameter/depth and skin/core temperatures will be taken from their CM prior to cooling the skin. The patients' CM will be cooled for a duration of 1 minute. The above measurements will be repeated immediately after 1 minute of cooling.

CONTACTS AND LOCATIONS:
Overall Officials: Irving Ling, MBBS, Principal Investigator — NHS Greater Glasgow and Clyde; Adam Gilmour, MBChB, MRCS (Ed), Study Chair — NHS Greater Glasgow and Clyde; Iain Mackay, MBChb, MRCS, FRCS (plast), Study Director — NHS Greater Glasgow and Clyde
Locations (1):
- Canniesburn Plastic Surgery Unit, Glasgow Royal Infirmary, Glasgow, United Kingdom